CLINICAL TRIAL: NCT04335019
Title: Interest of the Use of Pulmonary Ultrasound in the Referral of Patients With or Suspected COVID-19 +
Acronym: eChoVid
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200390; 2020-A00768-31 (Other: IDRCB)
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: 2019-nCoV (COVID-19); Interstitial Pneumonia
Keywords: Pulmonary ultrasound; Diagnosis improvement; Screening; 2019-nCoV (COVID-19); Chest CT
MeSH Terms: conditions — COVID-19; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pulmonary ultrasound — Pulmonary ultrasound results: quotation in 8 fields (right antero-superior, left antero-superior, right antero-inferior, left antero-inferior, right postero-superior, left postero-superior, right postero-inferior and postero-upper left).

SUMMARY:
The recent pandemic due to the SARS-CoV2 results in a pulmonary infection in major symptomatic patients. Because of the large number of patients and the risk of acute respiratory distress syndrome (which seems to occur in almost 5% of patients), there is a real challenge to improve physician ability to screen between patients those who will require specific surveillance and those who can be sent back home. The recent French official recommendation of the French radiology society prescribe that chest X-ray do not have any place in the COVID-19+ management whereas the WHO stipulate that ultrasound machines may be useful for these patients [1-2]. Moreover, scattered recent publications tend to stress the interest of quick ultrasound imaging for COVID-19 suspected patients for screening purpose [2-5].

The aim of this observational historico-prospective study is to assess the risk of severe clinical outcomes (admission in continuous care unit (USC), invasive respiratory assistance, death) in patients suspected or diagnosed COVID-19+ as a function of initial pulmonary ultrasound abnormalities. These clinical outcomes are assessed through phone calls at D5, D15, M1.

The secondary objectives are:

* Assessing the concordance between the severity of pulmonary lesions as detected by pulmonary ultrasound devices and the ones detected by CT-scanner, for patients who will undergo these two examinations.
* Assessing the compared performances in detecting ultrasound pulmonary lesions for patients suspected or diagnosed COVID-19+, between an experimented operator and a newly trained operator.
* Evaluate in suspected or COVID-19 patients, the risk of clinical worsening based on pulmonary ultrasound abnormalities during follow-up of hospitalized patients.
* Evaluate the ultrasound evolution profiles of pulmonary lesions in patients whose clinical evolution is favorable.
* Evaluate the incidence of thromboembolic events in patients who worsen secondarily.

DETAILED DESCRIPTION:
The practitioners involved at each site are

* either emergency physicians who are experts in pulmonary ultrasound
* either newly trained doctors who have received 30 minutes quick training in the fundamentals of pulmonary ultrasound.

The data collected under this protocol consists in:

* data from clinical examination: blood pressure, heart rate, respiratory rate, saturation, signs of confusion, body temperature, calculation of the CRB65 and qSOFA score, date of onset of symptoms
* Former patient journey: home, hospital, nursing home, others
* Medical background
* Recent use in the context of NSAID symptomatology
* Long-term use of nonsteroidal anti-inflammatory drugs (NSAIDs) in the context of a known pathology
* Results and date of PCR-Covid-19 test
* Pulmonary ultrasound results: quotation in 8 fields (right antero-superior, left antero-superior, right antero-inferior, left antero-inferior, right postero-superior, left postero-superior, right postero-inferior and postero-upper left).
* The operator's identity and level of expertise will be indicated.

Patients follow-up happens at D5, D15 and D28 through phone call. After verifying their identity using the initials entered and their date of birth, the patient or the referring person in the medical file is asked where the patient is currently (home, non ICU department, ICU department) and whether the patient is in respiratory assistance (invasive or not). In the event of notification of death, the date of occurrence will be indicated.

Patients are informed orally (in the event of altered state of consciousness, their close relative present will benefit from this information) that they will be contacted remotely (at D5, D15 and D28) to inquire about their development.

Patients hospitalized in most of the hospitals participating in the research will be offered a daily assessment of their clinical status, an ultrasound within 24-48 hours of the start of hospitalization, two other ultrasounds performed between D5 and D10. A final ultrasound will be performed before leaving the service.

In the event of worsening, a compression ultrasound of the lower limbs and a simple cardiac ultrasound is performed in search of signs of DVT or an acute pulmonary heart on a 4-point compression ultrasound and echocardiography which will be performed in the event of clinical worsening following the inclusion of the following :

* Evidence of a thrombus proximal to 4-point echo compression due to non-compressibility and / or absence of color doppler flow during a venous flushing maneuver
* Evidence of dilation of the ventricle Dt with VD / VG ratio> 1 or presence of a paradoxical septum.
* A search for the occurrence of one of these 3 events

  * Addressing in intensive care units
  * Mechanical ventilation
  * Death. In the event of notification of death, the date of occurrence will be indicated.

The report of the examination will be given on a standardized examination sheet with identification of the patient on each examination + identifier of the clinician operator.

The data will be kept for remote reading by a referent. All these examinations are carried out as part of the management of patients for the treatment of their COVID infection.

Patients are also informed:

* that any new information arising during the participation to the study, which could possibly modify his non opposition to this very participation, will be given
* of the right to have communication of information, held by the investigators, concerning their health, during or at the end of the research.
* Results of the chest scanner: typical COVID-19 and extent of the damage (minimal, moderate, severe)
* Initial patient orientation: return home, simple hospitalization or continuous care unit (USC), with or without respiratory assistance (and of what type: invasive or non-invasive), death (date of death)
* Whether or not to take chloroquine (on D0, D5, D15 or D28)
* Patient follow-up: same data as during the initial orientation on day 0, day 5, day 15 and D28.

ELIGIBILITY:
Inclusion criteria :

* > 18 years old
* Suspected of COVID-19 infection or having a systematic COVID-19 screening

Exclusion criteria :

* Patients on whom the ultrasonographic examination is not feasible for technical reasons (morbid obesity, thoracic extensive subcutaneous emphysema, absorbent subcutaneous infiltrations, ...)
* Patients with comorbidities justifying priority intensive care, not linked to the COVID-19 condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected of COVID-19 infection or having a systematic COVID-19 screening
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Association of pulmonary lesions on ultrasound on D0 classified according to three stages of severity | at day 0
  Association of pulmonary lesions on ultrasound on D0 classified according to three stages of severity
  * There are few B lines at the lung bases
  * Bi-lateralization of B lines, numerous diffuse and / or curtain sign
  * Presence of signs of pulmonary consolidation, hepatization of the lung and air bronchogram)

SECONDARY OUTCOMES:
Assessment of the agreement between a newly trained operator and an experienced operator of classification in one of the three stages of ultrasound gravity, by Cohen's kappa coefficient. | at day 0
  The operator's identity and level of expertise will be indicated:
  * emergency physicians who are experts in pulmonary ultrasound
  * newly trained doctors who have received 30 minutes quick training in the fundamentals of pulmonary ultrasound.
  Pulmonary ultrasound results:
  quotation in 8 fields (right antero-superior, left antero-superior, right antero-inferior, left antero-inferior, right postero-superior, left postero-superior, right postero-inferior and postero-upper left).
Estimate in patients who had a CT-scan on D0, the agreement in the evaluation of the severity of lung lesions via ultrasound vs. CT-scan, by Cohen's kappa coefficient | at day 0
  Pulmonary ultrasound results: quotation in 8 fields (right antero-superior, left antero-superior, right antero-inferior, left antero-inferior, right postero-superior, left postero-superior, right postero-inferior and postero-upper left).
  Results of the chest scanner: typical COVID-19 and extent of the damage (minimal, moderate, severe)
Measurement of the cumulative incidence of invasive mechanical ventilation | at day 5
  A search for the occurrence of one of these 3 events
  * Addressing in intensive care units
  * Mechanical ventilation
  * Death. In the event of notification of death, the date of occurrence will be indicated.
Measurement of survival | at day 5
  Patients follow-up happens at D5 through phone call. After verifying their identity using the initials entered and their date of birth, the patient or the referring person in the medical file is asked where the patient is currently (home, non ICU department, ICU department) and whether the patient is in respiratory assistance (invasive or not). In the event of notification of death, the date of occurrence will be indicated.
Measurement of the cumulative incidence of invasive mechanical ventilation | at day 15
  A search for the occurrence of one of these 3 events
  * Addressing in intensive care units
  * Mechanical ventilation
  * Death. In the event of notification of death, the date of occurrence will be indicated.
Measurement of survival | at day 15
  Patients follow-up happens at D15 through phone call. After verifying their identity using the initials entered and their date of birth, the patient or the referring person in the medical file is asked where the patient is currently (home, non ICU department, ICU department) and whether the patient is in respiratory assistance (invasive or not). In the event of notification of death, the date of occurrence will be indicated.
Measurement of the cumulative incidence of invasive mechanical ventilation | at day 28
  A search for the occurrence of one of these 3 events
  * Addressing in intensive care units
  * Mechanical ventilation
  * Death. In the event of notification of death, the date of occurrence will be indicated.
Measurement of survival | at day 28
  Patients follow-up happens at D28 through phone call. After verifying their identity using the initials entered and their date of birth, the patient or the referring person in the medical file is asked where the patient is currently (home, non ICU department, ICU department) and whether the patient is in respiratory assistance (invasive or not). In the event of notification of death, the date of occurrence will be indicated.
Association of the worsening of pulmonary lesions with the ultrasound | Within 48 hours of arrival in the service
  The kinetics of evolution of the pulmonary lesions with the favorable clinical evolution follow theses events:
  * stopping oxygen therapy
  * discharge from hospital
  * Presence of signs of DVT or an acute pulmonary heart on 4-point compression ultrasound and echocardiography
Association of the worsening of pulmonary lesions with the ultrasound | Between the 5th and 10 days of hospitalization
  The kinetics of evolution of the pulmonary lesions with the favorable clinical evolution follow theses events:
  * stopping oxygen therapy
  * discharge from hospital
  * Presence of signs of DVT or an acute pulmonary heart on 4-point compression ultrasound and echocardiography
Association of the worsening of pulmonary lesions with the ultrasound | just before discharge from hospital or in case of worsening
  The kinetics of evolution of the pulmonary lesions with the favorable clinical evolution follow theses events:
  * stopping oxygen therapy
  * discharge from hospital
  * Presence of signs of DVT or an acute pulmonary heart on 4-point compression ultrasound and echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi BENCHOUFI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Urgences - Hôpital Cochin APHP, Paris, France

REFERENCES:
- [Background] The recommendations of the French Radiology Society in the context of COVID-19 [Internet]. [cited 2020 Apr 1]. Available from: http://www.thema-radiologie.fr/actualites/2618/les-recommandations-de-la-societe-francaise-de-radiologie-dans-un-contexte-de-covid-19.html
- [Background] WHO | Disease Commodity Packages [Internet]. [cited 2020 Apr 1]. Available from: https://www.who.int/emergencies/what-we-do/prevention-readiness/disease-commodity-packages/en/
- [Background] Peng QY, Wang XT, Zhang LN; Chinese Critical Care Ultrasound Study Group (CCUSG). Findings of lung ultrasonography of novel corona virus pneumonia during the 2019-2020 epidemic. Intensive Care Med. 2020 May;46(5):849-850. doi: 10.1007/s00134-020-05996-6. Epub 2020 Mar 12. No abstract available. PMID 32166346
- [Background] Poggiali E, Dacrema A, Bastoni D, Tinelli V, Demichele E, Mateo Ramos P, Marciano T, Silva M, Vercelli A, Magnacavallo A. Can Lung US Help Critical Care Clinicians in the Early Diagnosis of Novel Coronavirus (COVID-19) Pneumonia? Radiology. 2020 Jun;295(3):E6. doi: 10.1148/radiol.2020200847. Epub 2020 Mar 13. No abstract available. PMID 32167853
- [Background] Buonsenso D, Pata D, Chiaretti A. COVID-19 outbreak: less stethoscope, more ultrasound. Lancet Respir Med. 2020 May;8(5):e27. doi: 10.1016/S2213-2600(20)30120-X. Epub 2020 Mar 20. No abstract available. PMID 32203708